CLINICAL TRIAL: NCT02195960
Title: Supplementation With Dietary Anthocyanins and Side Effects of Radiotherapy for Breast Cancer
Acronym: ATHENA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Maria Benedetta Donati, head laboratory, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Neuromed-ATH-EU2014
Record Dates: First submitted 2014-06-03; First posted 2014-07-21 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Toxicity Due to Radiotherapy
Keywords: skin toxicity, radiotherapy, antioxidants

STUDY DESIGN:
Intervention Model Description: Corn cobs-derived extracts of soluble anthocyanins given to breast cancer patients undergoing radiotherapy, to test prevention of skin toxicity.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, doctors, RT technicians, investigators and statisticians who participated or evaluated the study outcomes were blinded to the nature of the supplements. Anthocyanin and placebo stick packs and soluble granulated products were identical for organoleptic properties and coded as A and B by the producer. Only after completion of statistical analyses of trial results, blind codes were opened by the provider.
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): intake corn extract poor in anthocyanins: three daily stick packs containing water-soluble extract from corn cobs poor in anthocyanins
  Interventions: Dietary Supplement: Placebo
- intake anthocyanin-rich corn extract (Active Comparator): intake anthocyanin-rich corn extract: three daily stick packs containing water-soluble extract from high-anthocyanin rich corn cobs
  Interventions: Dietary Supplement: intake anthocyanin-rich corn extract

INTERVENTIONS:
Dietary Supplement: Placebo — intake corn extract poor in anthocyanins: three daily stick packs containing water-soluble extract from corn cobs poor in anthocyanins
  Arms: placebo
Dietary Supplement: intake anthocyanin-rich corn extract — intake anthocyanin-rich corn extract: three daily stick packs containing water-soluble extract from high-anthocyanin rich corn cobs
  Arms: intake anthocyanin-rich corn extract

SUMMARY:
Attention has been focused recently on the development of modalities that can protect healthy organs from the harmful effects of radiation applied during different cancer treatment schedules. As radiation-induced DNA damage involves oxidative stress, the protective role of antioxidants has been tested in different dietary studies. Previous experience by the collaborative team of the principal investigator and radiotherapists at the Catholic University of Campobasso has shown in a retrospective study that moderate wine consumption can reduce the side-effects of radiation therapy in patients with breast cancer. This effect was presumably due to the polyphenol non alcoholic fraction of wine, a finding in agreement with a cross-over intervention study in adult male volunteers, on protection by de-alcoholized red wine from ex vivo radiation-induced DNA damage.

The purpose of this clinical trial will be to test the impact of supplementation with anthocyanin-enriched food on the acute and medium-term side effects of radiotherapy in breast cancer patients, in a prospective study design. Therefore a double blind, randomised, placebo-controlled clinical trial will be organised by assigning patients with breast cancer scheduled for radiotherapy to a diet supplemented with an anthocyanin soluble extract.

DETAILED DESCRIPTION:
Detailed Description

1. Study Rationale:

   Attention has been focused recently on the development of modalities that can protect healthy organs from the harmful effects of radiation applied during different cancer treatment schedules. As radiation-induced DNA and cellular damage involve oxidative stress, the protective role of antioxidants will be tested on the toxic condition induced by radiotherapy in breast cancer treatment. Consumption of polyphenol-rich foods, such as fruits and vegetables, and beverages derived from plants, such as cocoa, red wine and tea, may represent a beneficial diet in terms of oxidative protection. Indeed, a retrospective study reports that that moderate wine consumption can reduce the side-effects of radiation therapy in patients with breast cancer. This effect was presumably due to the polyphenol non alcoholic fraction of wine, a finding in agreement with a cross-over intervention study in adult male volunteers, on protection by de-alcoholized red wine from ex vivo radiation-induced DNA damage. However, there are no studies that address the relationship of polyphenol-rich food consumption with the toxic effects of radiations in patients undergoing radiotherapy for breast cancer treatment.
2. Aim of the study. The main objectives of this study are to evaluate the association between the effect of polyphenol-rich food supplementation and toxicity of radiotherapy for breast cancer.
3. Study design: Randomized, placebo-controlled double-blind trial with 2 parallel arms: soluble corn flour at high content in anthocyanins and placebo. Placebo consists of soluble corn flour poor in anthocyanins. The treatment will start one week before starting radiotherapy, and continue during all radiotherapy treatment (of 3 or 5 weeks).
4. Study Population and recruitment: A total of 300 consecutive breast cancer patients eligible for radiotherapy. Participants will be identified at the Department of Radiotherapy of the Giovanni Paolo II Foundation of Campobasso.

Eligible subjects will be recruited at their first consultation and subsequently referred to the research investigators. The research staff in charge of the recruitment will pre-screen participants on the basis of inclusion/exclusion criteria and will explain the study at this time.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must consent to be in the study and must have signed an approved consent form conforming with institutional guidelines.
2. Patients must be ≥ 18 years old.
3. On histological examination, the tumor must be DCIS or invasive carcinoma of the breast.
4. Surgical treatment of the breast must have been lumpectomy or quadrantectomy. The margins of the resected specimen must be histologically free of tumor (DCIS and invasive). Reexcision of surgical margins is permitted.
5. Patients with invasive breast cancer are required to have axillary staging which can include sentinel node biopsy alone (if sentinel node is negative), sentinel node biopsy followed by axillary dissection or sampling with a minimum total of 6 axillary nodes (if sentinel node is positive), or axillary dissection alone (with a minimum of 6 axillary nodes). (Axillary staging is not required for patients with DCIS.)
6. The patient must be randomized within 45 days following the last surgery for breast cancer (lumpectomy, re-excision of margins, or axillary staging procedure) or within 30 days following the last chemotherapy cycle.
7. Patients with a history of non-breast malignancies are eligible if they have been disease-free for 5 or more years prior to randomization and are deemed by their physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.

Exclusion Criteria:

1. Axillary nodes with definite evidence of microscopic or macroscopic extracapsular extension.
2. One or more positive non-axillary sentinel node(s). (Note that intramammary nodes are staged as axillary nodes.)
3. Palpable or radiographically suspicious ipsilateral or contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes, unless there is histologic confirmation that these nodes are negative for tumor.
4. Suspicious microcalcifications, densities, or palpable abnormalities (in the ipsilateral or contralateral breast) unless biopsied and found to be benign.
5. Non-epithelial breast malignancies such as sarcoma or lymphoma.
6. Proven multicentric carcinoma (invasive cancer or DCIS) in more than one quadrant or separated by 4 or more centimeters.
7. Paget's disease of the nipple.
8. Synchronous bilateral invasive or non-invasive breast cancer.
9. Surgical margins that cannot be microscopically assessed or are positive at pathologic evaluation. (If surgical margins are rendered free of disease by reexcision, the patient is eligible.)
10. Breast implants. (Patients who have had implants removed are eligible.)
11. Prior breast or thoracic radiation therapy for any condition.
12. Collagen vascular disease, specifically dermatomyositis with a creatine phosphokinase level above normal or with an active skin rash, systemic lupus erythematosus, or scleroderma.
13. Pregnancy or lactation at the time of proposed randomization. Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy.
14. Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2014-06-09 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
side effects of radiotherapy | 4 or 6 weeks, according to the radiotherapy protocol
  Prevention of side effects - skin toxicity - of radiotherapy

SECONDARY OUTCOMES:
Acute skin toxicity | 1 month after the end of treatment (8 or 10 weeks)
  Secondary end-points are late toxicity, cosmetic results, local control, and survival.
Peripheral markers of inflammation | before starting treatment, at the end (4 or 6 weeks) and 1 month after radiotherapy (8 or 10 weeks)
  Blood cells count, markers of plasma and cell oxidation, markers of inflammatory response and oxidative DNA damage
Peripheral markers of bioavailability | before starting and at the end of treatment (4 or 6 weeks)
  Anthocyanins excretion will be evaluated in urine samples by analytical techniques.

OTHER OUTCOMES:
long-term skin toxicity | 6 and 12 months after the end of radiotherapy, corresponding to 7 or 7.5 months and 13 or 13.5 months from the beginning of the study
  late toxicity, cosmetic results, local control, and survival

CONTACTS AND LOCATIONS:
Overall Officials: Maria Benedetta Donati, MD PhD, Principal Investigator — Neuromed IRCCS
Locations (1):
- Department of Radiotherapy, Campobasso, CB, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bracone F, De Curtis A, Di Castelnuovo A, Pilu R, Boccardi M, Cilla S, Macchia G, Deodato F, Costanzo S, Iacoviello L, de Gaetano G, Morganti AG, Petroni K, Tonelli C, Donati MB, Cerletti C; EU-ATHENA Trial Investigators. Skin toxicity following radiotherapy in patients with breast carcinoma: is anthocyanin supplementation beneficial? Clin Nutr. 2021 Apr;40(4):2068-2077. doi: 10.1016/j.clnu.2020.09.030. Epub 2020 Oct 6. PMID 33051045